CLINICAL TRIAL: NCT01085591
Title: A Randomized, Double-Blinded, Active-Controlled, Dose Ranging Study of CB-183,315 in Patients With Clostridium Difficile Infection.
Brief Title: Study of CB-183,315 in Participants With Clostridium Difficile Infection
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Cubist Pharmaceuticals LLC, a subsidiary of Merck & Co., Inc. (Rahway, New Jersey USA) (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 4261-007; LCD-DR-09-03 (Other: Cubist Study Number)
Record Dates: First submitted 2010-03-09; First posted 2010-03-12 (Estimated); Results first posted 2015-06-16 (Estimated); Last update posted 2018-09-11 (Actual); Status verified 2018-08

CONDITIONS: Clostridium Difficile Infection; Diarrhea
Keywords: CDI; Clostridium difficile Infection; Diarrhea
MeSH Terms: conditions — Clostridium Infections; Diarrhea | interventions — CB-183,315; Vancomycin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- CB-183,315, 125 mg (Experimental): 125 milligrams (mg) CB 183,315 administered orally twice daily, alternating with twice daily oral administration of placebo tablets, for 10 days.
  Interventions: Drug: CB-183,315; Drug: Placebo
- CB-183,315, 250 mg (Experimental): 250 mg CB 183,315 administered orally twice daily, alternating with twice daily oral administration of placebo tablets, for 10 days.
  Interventions: Drug: CB-183,315; Drug: Placebo
- Vancomycin, 125 mg (Active Comparator): 125 mg vancomycin administered orally four times a day for 10 days.
  Interventions: Drug: Vancomycin

INTERVENTIONS:
Drug: CB-183,315
  Arms: CB-183,315, 125 mg; CB-183,315, 250 mg
Drug: Placebo
  Arms: CB-183,315, 125 mg; CB-183,315, 250 mg
Drug: Vancomycin
  Arms: Vancomycin, 125 mg

SUMMARY:
This is a randomized, double-blind, single-placebo, active-controlled, dose ranging parallel group design with 3 arms. Two dose regimens of CB-183,315 dosed twice daily will be compared with the active comparator oral vancomycin (125 milligrams (mg ) four times daily). Participants with diarrhea at risk for Clostridium difficile infection (CDI) [for example, received prior or concomitant antibiotic(s)] will be identified and tested for C. difficile toxin in stool using an enzyme immunoassay (EIA), or polymerase chain reaction (PCR) per the usual standard of care. Eligible participants will be consented, undergo baseline evaluations, and will be randomized in a blinded fashion to one of 3 treatment arms.

Participants will be randomized to receive either 125 mg CB-183,315 twice daily alternating with placebo tablets twice daily, 250 mg CB-183,315 twice daily alternating with placebo tablets twice daily or 125 mg oral vancomycin four times dailyover a period of 10 days in a 1:1:1 fashion.

ELIGIBILITY:
To be eligible for enrollment, a participant must meet all of the following criteria prior to any study related procedures:

* Informed Consent obtained and signed
* Age ≥ 18 years
* If female, participant is non-lactating, and is either:

  * Not of childbearing potential, defined as postmenopausal for at least 1 year or surgically sterile due to bilateral tubal ligation, bilateral oophorectomy, or hysterectomy
  * Of childbearing potential and is practicing the barrier method of birth control along with one of the following methods: oral or parenteral contraceptives for 3 months prior to study drug administration, a vasectomized partner, or abstinence from sexual intercourse
* Established non-severe or severe CDI (after Data Monitoring Committee [DMC] review) with a positive stool test for toxin A and/or B within 72 hours prior to first dose of study drug.

Exclusion Criteria:

A participant will not be enrolled if s/he meets any of the following criteria:

* Female and pregnant or lactating
* Toxic megacolon and/or known small bowel ileus
* Received treatment with intravenous (IV) immune globulin within 30 days prior to the first dose of study drug
* Antibacterial therapy specific for current CDI or that may be effective for CDI even if given for a different indication:

  * Received more than 24 hours of oral vancomycin for the current episode of CDI prior to first dose of study drug.
  * Received more than 24 hours of oral/intravenous metronidazole OR any other therapy specific for the current episode of CDI immediately prior to first dose of study drug unless the participant received at least 3 days of such therapy, and is considered a treatment failure for CDI.
  * Received more than 24 hours of oral/intravenous metronidazole for any other indication in the 3 days prior to first dose of study drug.
* Participants with more than 2 episodes of CDI within 90 days (that is, participants can be enrolled with their 1st recurrence/2nd episode)
* Major gastrointestinal (GI) surgery (that is, significant bowel resection including total colectomy with ileostomy) within 3 months of enrollment (this does not include appendectomy or cholecystectomy)
* History of prior inflammatory bowel disease: ulcerative colitis, Crohn's disease, or microscopic colitis
* Unable to stop loperamide, diphenoxylate, and cholestyramine during the duration of the study
* Unable to stop opiate treatment, unless on a stable dose as of onset of diarrhea and no change in dose planned for the duration of the study
* Known positive stool cultures for other enteropathogens, including but not limited to Salmonella, Shigella and Campylobacter
* Known stool studies positive for ova and/or parasites
* Known intolerance or hypersensitivity to daptomycin and/or vancomycin
* Poor concurrent medical risks with clinically significant co-morbid disease such that in the opinion of the Investigator the participant should not be enrolled
* Received an investigational drug or participated in any experimental procedure within 1 month prior to study entry
* Previously enrolled in this study
* Received an investigational vaccine against C. difficile
* Participants with known Hepatitis B or Hepatitis C who have alanine aminotransferase or aspartate aminotransferase > 2.5 times the upper limit of normal (ULN) and/or bilirubin > 1.5 times the ULN
* Human immunodeficiency virus positive, unless controlled (that is, on triple therapy) and with a CD4 > 200 cells per millimeter cubed (cellsmm˄3)
* Anticipated that systemic antibacterial therapy for a non-CDI infections will be required for >7 days after start of study therapy
* Concurrent therapy with daptomycin
* Unable to discontinue Saccharomyces or similar probiotic
* Known active IV drug or alcohol abuse
* Concurrent intensive chemotherapy, radiotherapy or biologic treatment for active malignancy (may only be enrolled after consultation with Medical Monitor)
* Unable to comply with the protocol requirements
* Any condition that, in the opinion of the Investigator, might interfere with study objectives
* Life expectancy is less than 6 weeks

Additional Exclusions for Participants with Severe CDI

In addition to the criteria listed above, a participant who meets the definition of severe CDI will not be enrolled if the participant meets any of the following criteria:

* Age > 80
* Hypotension, defined by sustained systolic blood pressure < 90 millimeters of mercury (mmHg), or need for vasopressors to maintain blood pressure
* Abdominal rebound tenderness on examination
* Acute kidney insufficiency defined by:

  * oliguria (< 20 cubic centimeter [cc] urine output per hour over a 4 hour period not responsive to attempts to increase renal perfusion) or
  * non-perfusion (for example, pre-renal) related azotemia with initial creatinine (Baseline) > 2.5 milligrams per deciliter (mg/dL) and blood urea nitrogen (BUN) > 40 mg/dL with no prior history of chronic kidney disease
* Unable to tolerate oral medications due to persistent vomiting 2. White blood cell (WBC) count > 30,000/mm˄3

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 210 (Actual)
Dates: Start 2010-04-01 (Actual); Primary Completion 2011-04-13 (Actual); Study Completion 2011-05-13 (Actual)

CONTACTS AND LOCATIONS:
Locations (32):
- United States (22):
  - Providence Hospital Clinical Research Center, Washington D.C., District of Columbia
  - Washington Hospital Center, Washington D.C., District of Columbia
  - Central Florida Internists, Saint Cloud, Florida
  - Atlanta Institute for Medical Research, Inc, Decatur, Georgia
  - Gastrointestinal Specialists of Georgia PC, Marietta, Georgia
  - Wellstar Infectious Disease, Marietta, Georgia
  - Idaho Falls Infectious Disease, PLLC, Idaho City, Idaho
  - University of Chicago, Chicago, Illinois
  - University of Kansas Medical Center, Kansas City, Kansas
  - Ochsner Clinic Foundation, New Orleans, Louisiana
  - Metropolitan Gastroentrology Group, Chevy Chase, Maryland
  - Tufts University School of Medicine, Boston, Massachusetts
  - Henry Ford Health System, Detroit, Michigan
  - Keego Harbor, Michigan
  - William Beaumont Hospital, Royal Oak, Michigan
  - University of Minnesota, Minneapolis, Minnesota
  - Missouri Baptist Medical Center, St Louis, Missouri
  - Mercury Street Medical Group - Research Group, Butte, Montana
  - DiGiovanna Institute for Medical Education and Research, North Massapequa, New York
  - Wake Forest University Health Sciences, Winston-Salem, North Carolina
  - MeritCare Clinical Research, Fargo, North Dakota
  - Remington Davis Inc., Columbus, Ohio
- Canada (10):
  - University of Calgary, Foothills Medical Center, Calgary, Alberta
  - St. Joseph Healthcare, Hamilton, Ontario
  - Queen's University, Kingston, Ontario
  - Mount Sinai Hospital, Toronto, Ontario
  - Centre de Sante et des Services Sociaux de Chicoutimi, Chicoutimi, Quebec
  - Maisonneuve Rosemont Hospital, Montreal, Quebec
  - SMBD- Jewish General Hospital G-139, Montreal, Quebec
  - Centre Hospitalier Universitaire de Québec, Québec, Quebec
  - Centre Hospitalier Universitaire de Sherbrooke, Sherbrook, Quebec
  - Centre hopitalier regional de Trois-Rivieres, Trois-Rivières, Quebec

IPD SHARING:
Plan to Share IPD: Yes
https://www.merck.com/clinical-trials/pdf/ProcedureAccessClinicalTrialData.pdf
URL: http://engagezone.msd.com/ds_documentation.php

REFERENCES:
- [Result] Lee CH, Patino H, Stevens C, Rege S, Chesnel L, Louie T, Mullane KM. Surotomycin versus vancomycin for Clostridium difficile infection: Phase 2, randomized, controlled, double-blind, non-inferiority, multicentre trial. J Antimicrob Chemother. 2016 Oct;71(10):2964-71. doi: 10.1093/jac/dkw246. Epub 2016 Jul 17. PMID 27432604

RESULTS

PARTICIPANT FLOW:
Groups:
- CB-183,315, 125 mg: 125 milligrams (mg) CB-183,315 administered orally twice daily, alternating with twice daily oral administration of placebo tablets, for 10 days
- CB-183,315, 250 mg: 250 mg CB-183,315 administered orally twice daily, alternating with twice daily oral administration of placebo tablets, for 10 days.
- Oral Vancomycin, 125 mg: 125 mg vancomycin administered orally four times a day for 10 days
Period: Overall Study
Arm/Group | CB-183,315, 125 mg | CB-183,315, 250 mg | Oral Vancomycin, 125 mg
Started | 69 | 71 | 70
Received at Least 1 Dose of Study Drug | 68 | 69 | 70
Completed | 66 | 65 | 63
Not Completed | 3 | 6 | 7
Not completed — Adverse Event | 0 | 1 | 3
Not completed — Physician Decision | 1 | 0 | 1
Not completed — Withdrawal by Subject | 0 | 2 | 1
Not completed — Lost to Follow-up | 0 | 1 | 1
Not completed — Protocol Violation | 1 | 1 | 1
Not completed — Other | 0 | 1 | 0
Not completed — Not Properly Consented | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Population: All randomized participants who gave proper informed consent.
Groups:
- Total: Total of all reporting groups
Arm/Group | CB-183,315, 125 mg | CB-183,315, 250 mg | Oral Vancomycin, 125 mg | Total
Number analyzed (Participants) | 68 | 71 | 70 | 209
Age, Categorical [Count of Participants; unit: Participants]
  LTE18 | 0 | 0 | 0 | 0
  BTWN | 47 | 43 | 40 | 130
  GTE65 | 21 | 28 | 30 | 79
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 45 | 43 | 44 | 132
  Male | 23 | 28 | 26 | 77

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With a Clinical Response Outcome of Clostridium Difficile Infection Cure at the End of Study Treatment
Description: The number of participants with an Investigator-assessed clinical response of cure is presented. The information to assess clinical response was collected at any time up to and including Day 19.
Time Frame: Baseline (Day 0) through Study Day 19
Population: All participants who received any amount of study drug and had a confirmed diagnosis of Clostridium difficile infection (CDI).
Measure: Number; unit: participants
Groups:
- CB-183,315, 125mg: 125 milligrams (mg) CB-183,315 administered orally twice daily, alternating with twice daily oral administration of placebo tablets, for 10 days
Arm/Group | CB-183,315, 125mg | CB-183,315, 250 mg | Oral Vancomycin, 125 mg
Number analyzed (Participants) | 66 | 67 | 66
participants | 61 | 58 | 59

2. Secondary Outcome: Number of Participants With a Recurrence of Clostridium Difficile Infection Through the 4-week Follow-up Period
Description: The number of participants with a recurrence of CDI is presented along with the number of participants without a recurrence and who were unable to be evaluated. Participants with a favorable outcome at the EOT (cure) were evaluated for recurrence of CDI. Only subjects deemed a cure at EOT were assessed for recurrence. This is the denominator used for all percentages. If diarrheal symptoms returned, participants were asked to indicate the number of unformed bowel movements (UBM) they had and have an additional C. difficile toxin test. The information to assess recurrence in participants who were deemed a cure at EOT was collected at any time during the 4-week Follow-up Period (FUP).
Time Frame: Study Day 10 up to Study Day 40
Population: as for outcome 1
Measure: Number; unit: Participants
Arm/Group | CB-183,315, 125 mg | CB-183,315, 250 mg | Oral Vancomycin, 125 mg
Number analyzed (Participants) | 61 | 58 | 59
Participants
  Recurrence of CDI | 17 | 10 | 21
  No Recurrence of CDI | 44 | 47 | 37
  Unable to Evaluate | 0 | 1 | 1

3. Secondary Outcome: Number of Participants With a Clinical Response Outcome at the End of Study Treatment With and Without Infection Caused by C. Difficile BI/NAP1/027 Strain at Baseline
Description: The number of participants with investigator assessed clinical response of cure, failure or unable to evaluate is presented and shown separately for participants with and without infection caused by C. difficile BI/NAP1/027 strain as determined at baseline. Clinical response was determined by the participant's condition on the second day following the last dose of study medication, unless considered a treatment failure. Treatment failures were assessed whenever they occurred and were carried forward to the EOT. The information to assess clinical response for infection caused by C. difficile BI/NAP1/027 strain at Baseline was collected at any time up to and including Day 12. Strain at Baseline=SAB
Time Frame: Baseline (Day 0) through Study Day 12
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | CB-183,315, 125 mg | CB-183,315, 250 mg | Oral Vancomycin, 125 mg
Number analyzed (Participants) | 66 | 67 | 66
participants
  Cure of CDI with BI/NAP1/027 SAB (n=18, 21, 23) | 15 | 15 | 21
  Failure with SAB (n=18, 21, 23) | 1 | 4 | 1
  Unable to Evaluate with SAB (n=18, 21, 23) | 2 | 2 | 1
  Cure of CDI without SAB (n=44, 37, 38) | 42 | 34 | 34
  Failure without SAB (n=44, 37, 38) | 2 | 1 | 2
  Unable to Evaluate without SAB (n=44, 37, 38) | 0 | 2 | 2

4. Secondary Outcome: Number of Participants With a Recurrence of Clostridium Difficile Infection at the End of Study Treatment With and Without Infection Caused by C. Difficile BI/NAP1/027 Strain at Baseline
Description: The number of participants with and without infection caused by C. difficile BI/NAP1/027 strain as determined at baseline with a recurrence of CDI is presented along with the number of participants without a recurrence and who were unable to be evaluated. Participants with a favorable outcome at the EOT (cure) were evaluated for recurrence of CDI. If diarrheal symptoms returned, participants were asked to indicate the number of UBM they had and have an additional C. difficile toxin test. The information to assess recurrence in participants who were deemed a cure at EOT was collected at any time during the 4-week FUP. Strain at Baseline=SAB.
Time Frame: Study Day 10 up to Study Day 40
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | CB-183,315, 125 mg | CB-183,315, 250 mg | Oral Vancomycin, 125 mg
Number analyzed (Participants) | 66 | 67 | 66
participants
  Recurrence of CDI with SAB (n=15, 15, 21) | 5 | 5 | 11
  No Recurrence of CDI with SAB (n=15,15, 21) | 10 | 9 | 10
  Unable to Evaluate with SAB (n=15,15, 21) | 0 | 1 | 0
  Recurrence of CDI without SAB (n=42, 34, 34) | 11 | 5 | 8
  No Recurrence of CDI without SAB (n=42, 34, 34) | 31 | 29 | 25
  Unable to Evaluate without SAB (n=42, 34, 34) | 0 | 0 | 1

5. Secondary Outcome: Median Time to Resolution of Diarrhea
Description: The median time to resolution of diarrhea is presented for evaluable participants in each treatment group. The time in days from the start of treatment (time of first dose of study drug) to resolution (time of the last UBM on the day before the first of 2 consecutive days of < 4 UBMs and sustained through the second day following the last dose of study drug).
Time Frame: Baseline (Day 0) through Study Day 12
Population: All participants who received any amount of study drug, had a confirmed diagnosis of Clostridium difficile infection (CDI), and who achieved resolution of their diarrhea.
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | CB-183,315, 125 mg | CB-183,315, 250 mg | Oral Vancomycin, 125 mg
Number analyzed (Participants) | 58 | 57 | 56
Days | 1.5 [0.6 to 2.40] | 1.4 [0.90 to 2.30] | 2.1 [1.40 to 2.50]

6. Primary Outcome: Number of Participants With a Clinical Response Outcome of Failure or Unable to Evaluate at the End of Study Treatment
Description: The number of participants with investigator assessed clinical response of failure or unable to evaluate is presented. Clinical response was determined by the participant's condition on the second day following the last dose of study medication, unless considered a treatment failure. Treatment failures were assessed whenever they occurred and were carried forward to the end-of-treatment (EOT). The information to assess clinical response was collected at any time up to and including Day 19.
Time Frame: Baseline (Day 0) through Study Day 19
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | CB-183,315, 125 mg | CB-183,315, 250 mg | Oral Vancomycin, 125 mg
Number analyzed (Participants) | 66 | 67 | 66
participants
  Failure | 3 | 5 | 4
  Unable to Evaluate | 2 | 4 | 3

ADVERSE EVENTS:
Arm/Group | CB-183,315, 125 mg | CB-183,315, 250 mg | Oral Vancomycin, 125 mg
Serious Adverse Events (participants affected / at risk) | 12/68 | 6/69 | 11/70
Other Adverse Events (participants affected / at risk) | 34/68 | 43/69 | 41/70
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | CB-183,315, 125 mg (N=68) | CB-183,315, 250 mg (N=69) | Oral Vancomycin, 125 mg (N=70)
Cardiac arrest (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) — This SAE led to death for one participant in the oral vancomycin treatment group. Death occurred on day of last dose (fourth day of treatment)
Hypoacusis (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 1 (1) | 1 (1)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (2) — This SAE led to death for one participant in the CB-183,315 125mg treatment group. Death occurred 29 days after last dose
Peritonitis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Asthenia (General disorders) | 1 (1) | 0 (0) | 0 (0)
Graft versus host disease (Immune system disorders) | 1 (1) | 0 (0) | 0 (0)
Clostridial infection (Infections and infestations) | 4 (4) | 3 (3) | 4 (4)
Cytomegalovirus infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Endocarditis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 1 (1) | 0 (0) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Breast cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) — This SAE led to death for one participant in the CB-183,315 250mg treatment group. Death occurred 15 days after last dose
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) — This SAE led to death for one participant in the oral vancomycin treatment group. Death occurred 10 days after last dose
Haematuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
Renal failure acute (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Arterial thrombosis (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | CB-183,315, 125 mg (N=68) | CB-183,315, 250 mg (N=69) | Oral Vancomycin, 125 mg (N=70)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 1 (1)
Heparin-induced thrombocytopenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0)
Leukocytosis (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1)
Lymphadenopathy (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0)
Pancytopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1)
Cardiac failure congestive (Cardiac disorders) | 0 (0) | 1 (1) | 1 (1)
Palpitations (Cardiac disorders) | 1 (1) | 1 (1) | 2 (2)
Tachycardia (Cardiac disorders) | 1 (1) | 1 (1) | 1 (1)
Ear pain (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 0 (0)
Hypoacusis (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 1 (1)
Inner ear inflammation (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 1 (1)
Tinnitus (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 1 (1)
Tympanic membrane disorder (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 0 (0)
Conjunctival discolouration (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
Conjunctival haemorrhage (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
Photophobia (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
Vision blurred (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
Abdominal discomfort (Gastrointestinal disorders) | 1 (1) | 1 (1) | 1 (1)
Abdominal distension (Gastrointestinal disorders) | 2 (2) | 2 (2) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 3 (3) | 4 (5) | 7 (9)
Abdominal pain lower (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Abdominal pain upper (Gastrointestinal disorders) | 2 (2) | 0 (0) | 2 (2)
Abdominal tenderness (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Anal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Anorectal discomfort (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Constipation (Gastrointestinal disorders) | 1 (1) | 2 (2) | 1 (2)
Diarrhoea (Gastrointestinal disorders) | 3 (3) | 2 (2) | 2 (2)
Dry mouth (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 1 (1) | 3 (3) | 1 (1)
Dysphagia (Gastrointestinal disorders) | 0 (0) | 3 (3) | 1 (1)
Eructation (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Faecal incontinence (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Flatulence (Gastrointestinal disorders) | 3 (3) | 2 (2) | 5 (5)
Food poisoning (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Haematochezia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Haemorrhoids (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0)
Ileus (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Intestinal ischaemia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Melaena (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 8 (9) | 8 (9) | 4 (5)
Paraesthesia oral (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Rectal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1)
Rectal tenesmus (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 3 (4) | 1 (1) | 2 (3)
Asthenia (General disorders) | 1 (1) | 0 (0) | 3 (3)
Chest discomfort (General disorders) | 0 (0) | 0 (0) | 1 (1)
Chest pain (General disorders) | 1 (1) | 1 (1) | 0 (0)
Chills (General disorders) | 1 (1) | 1 (1) | 1 (1)
Dysplasia (General disorders) | 0 (0) | 1 (1) | 0 (0)
Fatigue (General disorders) | 4 (4) | 5 (6) | 4 (4)
Feeling abnormal (General disorders) | 0 (0) | 0 (0) | 1 (1)
Feeling hot (General disorders) | 0 (0) | 1 (1) | 0 (0)
Hyperthermia (General disorders) | 0 (0) | 1 (1) | 0 (0)
Inflammation (General disorders) | 0 (0) | 1 (1) | 0 (0)
Infusion site erythema (General disorders) | 0 (0) | 0 (0) | 1 (1)
Injection site haematoma (General disorders) | 1 (1) | 0 (0) | 0 (0)
Oedema (General disorders) | 0 (0) | 1 (1) | 0 (0)
Oedema peripheral (General disorders) | 1 (1) | 3 (3) | 2 (3)
Pelvic mass (General disorders) | 0 (0) | 0 (0) | 1 (1)
Pyrexia (General disorders) | 3 (3) | 1 (1) | 0 (0)
Tenderness (General disorders) | 2 (2) | 0 (0) | 0 (0)
Drug hypersensitivity (Immune system disorders) | 0 (0) | 1 (1) | 0 (0)
Acarodermatitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Candidiasis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Candiduria (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Enterococcal infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Fungal skin infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Gastroenteritis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Gastroenteritis viral (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Hordeolum (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Incision site infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Injection site infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Nasopharyngitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Oral candidiasis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Oral herpes (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Otitis externa (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Pharyngitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 3 (3)
Tinea cruris (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 1 (1) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 1 (1) | 4 (4) | 4 (4)
Vulvovaginal mycotic infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Accidental overdose (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 2 (3) | 1 (1) | 1 (1)
Head injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Joint dislocation (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Joint sprain (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Rib fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Sunburn (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Therapeutic agent toxicity (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Wound (Injury, poisoning and procedural complications) | 0 (0) | 2 (2) | 0 (0)
Alanine aminotransferase increased (Investigations) | 1 (1) | 1 (1) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 1 (1) | 1 (1) | 0 (0)
Bilirubin conjugated increased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Blood bilirubin unconjugated increased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Blood creatine phosphokinase increased (Investigations) | 3 (3) | 1 (1) | 1 (1)
Blood glucose abnormal (Investigations) | 0 (0) | 1 (1) | 0 (0)
Blood potassium decreased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Blood sodium decreased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Body temperature fluctuation (Investigations) | 0 (0) | 1 (1) | 0 (0)
Eosinophil count increased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Haemoglobin decreased (Investigations) | 1 (1) | 0 (0) | 0 (0)
International normalised ratio increased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Liver function test abnormal (Investigations) | 2 (2) | 0 (0) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 2 (2) | 3 (3) | 1 (1)
Gout (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Hyperkalaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Hypomagnesaemia (Metabolism and nutrition disorders) | 2 (2) | 1 (1) | 1 (1)
Hypophosphataemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Increased appetite (Metabolism and nutrition disorders) | 2 (2) | 0 (0) | 0 (0)
Malnutrition (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 3 (3)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 3 (3) | 0 (0)
Joint effusion (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Limb discomfort (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 1 (1)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 1 (1)
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2) | 0 (0)
Neck pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0) | 1 (1)
Carpal tunnel syndrome (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 2 (2) | 1 (1) | 5 (5)
Dysgeusia (Nervous system disorders) | 1 (1) | 1 (1) | 3 (3)
Headache (Nervous system disorders) | 6 (8) | 8 (14) | 3 (4)
Memory impairment (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Paraesthesia (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1)
Tremor (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Agitation (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
Anxiety (Psychiatric disorders) | 0 (0) | 1 (1) | 1 (1)
Depressed mood (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
Depression (Psychiatric disorders) | 1 (1) | 1 (1) | 0 (0)
Drug dependence (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
Insomnia (Psychiatric disorders) | 0 (0) | 1 (1) | 1 (1)
Dysuria (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Haematuria (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Oliguria (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Pollakiuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
Urinary incontinence (Renal and urinary disorders) | 1 (1) | 2 (2) | 0 (0)
Dysmenorrhoea (Reproductive system and breast disorders) | 0/45 (0) | 0/41 (0) | 1/44 (1)
Menstrual disorder (Reproductive system and breast disorders) | 0/45 (0) | 1/41 (1) | 0/44 (0)
Vaginal haemorrhage (Reproductive system and breast disorders) | 1/45 (1) | 0/41 (0) | 1/44 (1)
Vulvovaginal pruritus (Reproductive system and breast disorders) | 0/45 (0) | 1/41 (1) | 0/44 (0)
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Hypoventilation (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Nasal dryness (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1)
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0 (0)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Yawning (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Alopecia (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Cold sweat (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 1 (1)
Ecchymosis (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (2) | 2 (2)
Erythema (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (2) | 1 (1)
Night sweats (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Onychoclasis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 2 (2)
Pruritus generalised (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Skin lesion (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Wound drainage (Surgical and medical procedures) | 1 (1) | 0 (0) | 0 (0)
Arterial thrombosis (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)
Embolism (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Hot flush (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)
Hypotension (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other